CLINICAL TRIAL: NCT01905319
Title: Juvenile Idiopathic Arthritis in Children in Estonia - an Epidemiological and Clinical Investigation.
Brief Title: Juvenile Idiopathic Arthritis in Children in Estonia.
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Chris Pruunsild, MD, PhD, University of Tartu
Other Study IDs: TARLA 0475;DARLA 0500
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Epidemiology
Keywords: juvenile idiopathic arthritis; incidence rate
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subsequent new juvenile arthritis cases: During years 1998-2000, all new subsequent cases of juvenile idiopathic arthritis diagnosed in Estonia were included in the study group.
  Interventions: Other: Blood collecting for storage of samples

INTERVENTIONS:
Other: Blood collecting for storage of samples

SUMMARY:
Aims of the study:

* to study the incidence rate of juvenile idiopathic arthritis (JIA) and it's clinical subtypes in Estonia for the years 1998-2000;
* to examine the course and short-term clinical outcome of JIA.

Method: a prospective population-based study carried on in 14 counties of Estonia

ELIGIBILITY:
Inclusion Criteria:

* The International League of Associations for Rheumatology (ILAR) criteria for juvenile idiopathic arthritis
* children aged 0-15 years who had arthritis of an unknown cause for at least six weeks with an onset of the disease during the study period

Exclusion Criteria:

* Children with infectious arthritis, postinfectious arthritis, traumatic arthritis and systemic connective tissue diseases

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: During years 1998-2000, 162 newly-diagnosed juvenile idiopathic arthritis cases from 14 counties of Estonia, were included to the study, among them 76 boys and 86 girls.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 1998-01; Primary Completion 2000-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Mean annual incidence rate of juvenile idiopathic arthritis in Estonia during years 1998-2000. | 3 years

REFERENCES:
- [Derived] Pullerits R, Schierbeck H, Uibo K, Liivamagi H, Tarraste S, Talvik T, Sundberg E, Pruunsild C. High mobility group box protein 1-A prognostic marker for structural joint damage in 10-year follow-up of patients with juvenile idiopathic arthritis. Semin Arthritis Rheum. 2017 Feb;46(4):444-450. doi: 10.1016/j.semarthrit.2016.08.017. Epub 2016 Aug 26. PMID 27756498